CLINICAL TRIAL: NCT04848636
Title: Sodium Assessment of the Cardiac Tissue in Chronic Kidney Disease Patients Using Sodium Magnetic Resonance Imaging
Brief Title: Cardiac Tissue Sodium Assessment in CKD Patients Using Sodium MRI
Status: Recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Chris McIntyre, Director of Kidney Clinical Research Unit, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 118891
Record Dates: First submitted 2021-03-31; First posted 2021-04-19 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Chronic Kidney Diseases; Dialysis; Complications; Sodium Retention
Keywords: Sodium MRI; Chronic Kidney Disease; Hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypernatremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Complete blood count, kidney function (serum creatinine, cystatin C for healthy controls and CKD patients, urea, and electrolytes), liver function, serum albumin, cardiac biomarkers (high-sensitivity cardiac Troponin T), C-reactive protein, serum glucose.
  A spot urine sample will be collected on the day of the study and will be analyzed for sodium, creatinine, protein, and albumin levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Controls: * Age greater than or equal to 18 years
  * lack of kidney disease, cardiovascular disease, diabetes, liver cirrhosis and peripheral edema
  Interventions: Diagnostic Test: Cardiac Sodium and Proton MRI
- Chronic Kidney Disease Patients: * Age greater than or equal to 18 years
  * evidence of kidney disease persisting > 3 months and no indications to start dialysis
  Interventions: Diagnostic Test: Cardiac Sodium and Proton MRI
- Hemodialysis Patients: * Age greater than or equal to 18 years
  * more than 3 months duration of therapy
  Interventions: Diagnostic Test: Cardiac Sodium and Proton MRI

INTERVENTIONS:
Diagnostic Test: Cardiac Sodium and Proton MRI — Sodium-23 MRI of the Heart Proton MRI of the Heart

SUMMARY:
Chronic kidney disease (CKD) is prevalent worldwide and affects around 10% of people living in developed health economies. As the kidney loses its function in patients with CKD, the kidneys are unable to filter toxins out of the blood as efficiently as those of healthy individuals. Arguably, sodium (salt) is the most relevant toxin in CKD and can build up in the kidneys of patients with CKD. Salt build-up has also been found to occur in the heart muscle tissue and could drive the development of scarring of the heart muscle tissue which contributes to heart failure.

Using sodium magnetic resonance imaging (MRI), we would like to measure the levels of salt in the heart muscle tissue. We will examine whether the heart muscle tissue has high salt levels, and if so, whether this relates to any heart defects. A conventional proton MRI will be done to measure heart function. The MRI images of healthy volunteers, CKD patients, and those on hemodialysis will be analyzed for levels of salt and the findings will then be compared to the cardiac biomarkers (proteins or enzymes that are released into the blood when the heart is damaged or stressed) and fibrosis (scarring) measured from each patient's proton MRI images to establish a possible correlation. This research has the potential to precede additional studies that may investigate the effect of diuretics (a drug that increases the production of urine) on the heart muscle tissue of CKD patients.

Using sodium magnetic resonance imaging (MRI), it is possible to measure the sodium content in the cardiac tissue of patients with kidney disease. In this research study, it will be investigated whether the elevated levels of sodium in patients with kidney disease is also present in their hearts, and if so, whether this relates to cardiac abnormalities. Cardiac sodium MRI images of healthy volunteers, hemodialysis patients, and CKD patients will be analyzed for sodium content. This sodium information will then be compared to the biomarkers of cardiac function and fibrosis measured from each patient's proton MRI images in order to establish a possible correlation. This research has the potential to precede additional studies that may investigate the effect of diuretics on the cardiac tissue of kidney disease patients.

DETAILED DESCRIPTION:
This study is a pilot exploratory study (preliminary project to assess the use of a heart sodium coil across a wide spectrum of kidney disease). We will recruit up to 150 participants: approximately 50 hemodialysis patients, 50 patients with various stages of chronic kidney disease, and 50 age and sex matched healthy participants to compare clinical characteristics to. This study involves one study visit at the Robarts Research Institute, London, Ontario lasting approximately 3 hours.

This study entails one visit where all participants will undergo a proton and sodium MRI scan of the heart. Prior to the scan, all participants will have their sitting blood pressure and heart rate measured three times consecutively using a standard automatic blood pressure monitor. In addition to this, all patient participants will have blood work collected, provide a spot urine sample, complete a salt intake questionnaire, and have their fluid volume measured using bioimpedance spectroscopy. Only those patients on hemodialysis will answer a single Time to Recovery Question in addition to the above.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* For patients on maintenance hemodialysis: more than 3 months duration of therapy
* For patients with CKD: evidence of kidney disease persisting > 3 months and no indications to start dialysis
* For healthy controls: lack of kidney disease, cardiovascular disease, diabetes, liver cirrhosis and peripheral edema

Exclusion Criteria:

* Pregnant, breastfeeding or intending pregnancy
* Contraindication to MRI scan

  * Inability to tolerate MRI due to patient size and/or known history of claustrophobia.
  * Mechanically implanted, electrically, or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, tattoos, shunt, surgical staples (including clips or metallic sutures and/or ear implants.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient participants with chronic kidney disease or currently receiving hemodialysis treatment from London Health Sciences Centre Regional Renal Program, London, Ontario
  Age and sex matched healthy participants
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-07-10 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in Cardiac Sodium Signal | Baseline
  Difference in Cardiac Sodium Signal between hemodialysis patients, chronic kidney disease patients, and sex and age-matched healthy adult controls.

SECONDARY OUTCOMES:
Dialysate Composition | Baseline
  Correlation between Cardiac Sodium Signal and dialysate composition.
Serum Sodium Concentration | Baseline
  Correlation between Cardiac Sodium Signal and serum sodium concentration. Serum sodium concentration will be measured from a blood sample in mmol/L.
Proton MRI Biomarkers | Baseline
  Correlation between Cardiac Sodium Signal and left ventricular mass, end diastolic volume, and left atrial volume.
T1 Mapping | Baseline
  Correlation between Cardiac Sodium Signal and T1 times in the left ventricular wall.
T2 Mapping | Baseline
  Correlation between Cardiac Sodium Signal and T2 times in the left ventricular wall.
Serum Albumin | Baseline
  Correlation between Cardiac Sodium Signal and serum albumin. Serum albumin will be measured from a blood sample in g/L.
Serum High-Sensitivity Troponin T | Baseline
  Correlation between Cardiac Sodium Signal and serum high-sensitivity troponin T. Serum high-sensitivity troponin T will be measured from a blood sample in ng/L.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W McIntyre, MD/PhD, Principal Investigator — London Health Sciences Centre - Victoria Hospital
Locations (1):
- Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No